CLINICAL TRIAL: NCT04893512
Title: First-In-Human Study Of Orally Administered CoV2-OGEN1 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: US Specialty Formulations, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CoV2-OGEN1-101
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orally administered CoV2-OGEN1- 2 dose schedule (Experimental): 50mcg,100mcg and 200mcg will be tested as single oral dose on day 1 and day 15. The dose will be in the form of oral suspension.
  Interventions: Drug: Orally Suspension of CoV2-OGEN1

INTERVENTIONS:
Drug: Orally Suspension of CoV2-OGEN1 — CoV2-OGEN1 will be supplied as a 10mL oral suspension in a plastic bottle containing 50-200 mcg of formulated drug

SUMMARY:
To evaluate the safety of 2 dose vaccination schedule of orally administered CoV2-OGEN1 In healthy subjects

DETAILED DESCRIPTION:
The study will be conducted at 1 site in NZ. Patients who sign an Informed Consent and meet all eligibility criteria will be administered oral doses of 50mcg, 100mcg and 200mcg CoV2-OGEN1 on Day 1 and Day 15 during Cohort 1-3 respectively . Follow up visit in all the 3 cohorts will be performed at 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 3 months, 6 months, and 12 months. One sentinel subject will be dosed at the start of each cohort and will be monitored for 24 hours post administration before the remainder of the cohort can be recruited. Each cohort will include one sentinel subject.

Dose escalation will be done after assessing all adverse events and their relatedness in atleast 9 participants out of 15 receiving Cov2-OGEN1 who have completed their week 6 FU visit.

In case three (3) or more participants receiving CoV2-OGEN1 withdraw before Visit 6 (Week 4) follow up visit, the dose escalation safety assessment will be made by assessing all Adverse Events and their relatedness status in all participants receiving CoV2-OGEN1 of the current Cohort.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfil all of the following criteria to be eligible for the study:

1. Capable of giving personal signed informed consent, which includes compliance with the requirements and restrictions listed in this protocol and be available for all study visits.
2. Must agree to collection of nasal wash, oral rinse, and venous blood per protocol and agree to have samples stored for secondary research.
3. Male or non-pregnant female, >/= to 18 years and </= 56 years of age at time of enrollment.
4. Body Mass Index (BMI) 18-35 kg/m^2 at screening.
5. Women of childbearing potential must agree to use or have practiced true abstinence or use at least one acceptable primary form of contraception. Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement).
6. Male subjects of childbearing potential: use of condoms to ensure effective contraception with a female partner of childbearing potential from first vaccination until 90 days after the last vaccination.
7. Male subjects agree to refrain from sperm donation from the time of first vaccination until 90 days after the last vaccination.
8. In good health as determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of subjects. (Note: Chronic medical diagnoses/conditions/medications should be stable for the last 60 days (no hospitalizations, emergency room (ER), or urgent care for condition or need for supplemental oxygen)).
9. Oral temperature is less than 100.0 degrees Fahrenheit (37.8 degrees Celsius).
10. Pulse no greater than 100 beats per minute.
11. Systolic blood pressure (BP) is 85 to 150 mm Hg, inclusive.
12. Clinical screening laboratory evaluations (Basic Metabolic Panel, White blood cell (WBC), Hemoglobin (Hgb), Hematocrit (HCT), RBC count, Mean Corpuscular Volume (MCV), Mean Corpuscular Hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC), platelets (PLTs), Total Neutrophils - Absolute (NEUT#), Eosinophils - Absolute (EO#), Monocytes - Absolute (MONO#), Basophils - Absolute (BASO#), Lymphocytes - Absolute (LYMPH#), alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), total bilirubin (T. Bili), Lipase, prothrombin time (PT), and partial thromboplastin time (PTT)) are within the acceptable normal reference ranges of the clinical laboratory. Subjects with out of range values may be included if the clinical laboratory or PI deem the out of range value to be clinically insignificant.
13. The subject must agree to refrain from donating blood or plasma during the study (outside of this study).

Exclusion criteria

Participants will be excluded from participation in the study if any of the following criteria are met at screening:

1. Positive pregnancy test either at screening or just prior to the first vaccine administration.
2. Participants who is breastfeeding or planning on breastfeeding from the time of the first vaccination through 60 days after the last vaccination.
3. Has any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation.
4. Acute or chronic gastrointestinal conditions such as Crohn's, Ulcerative Colitis, gastritis, proctitis, IBS, or any other inflammatory bowel disease.
5. Currently taking Histamine-2 (H2) Blocker, Proton Pump Inhibitor (PPI), Promotility Agent, or any chronic antacids.
6. Presence of self-reported or medically documented significant medical or psychiatric condition(s).
7. Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), uncontrolled hypertension, history of myocarditis or pericarditis as an adult, myocardial infarction (MI) within past 6 months, coronary artery bypass surgery or stent placement, or uncontrolled cardiac arrhythmia.
8. Neurological or neurodevelopmental conditions (e.g., history of migraines in the past 5 years, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease).
9. Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
10. Active autoimmune disease or any history of autoimmune disease determined by hx or lab/physical examination.
11. Individuals at high risk for severe COVID-19, including those with any of the following risk factors:

    1. T2DM
    2. Asthma
    3. Respiratory conditions (including emphysema or COPD)
    4. Tobacco use (vaping, smoking, chew) within 1 year
12. Chronic kidney disease, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2.
13. Immunocompromised individuals with known or suspected immunodeficiency, as determined by medical history or lab/physical examination.
14. Acute illness, as determined by the site PI or appropriate sub-investigator, with or without fever [oral temperature >/= 38.0 degrees Celsius (100.4 degrees Fahrenheit)] within 72 hours prior to each vaccination.
15. History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
16. Participation in another investigational study involving any investigational product within 60 days, or 5 half-lives, whichever is longer, before the first vaccine administration.
17. Participation in another clinical trial with an investigational agent that will be received during the study-reporting period.
18. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines.
19. Chronic use (more than 14 continuous days) or anticipated use within the next 6 months of any medications that may be associated with impaired immune responsiveness. Including, but not limited to the following excluded drugs: systemic or inhaled corticosteroids, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1). The use of low dose topical, ophthalmic, otic, and intranasal steroid preparations will be permitted.
20. Anticipating the need for immunosuppressive treatment within the next 6 months.
21. Receipt of immunoglobulin and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
22. Blood dyscrasias or significant disorder of coagulation, based on history or abnormal laboratory results.
23. Chronic liver disease, including fatty liver.
24. Has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 6 months before the first vaccine administration.
25. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
26. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
27. Receipt of any other SARS-CoV-2, MERS, SARS-CoV-1 or other experimental coronavirus vaccine at any time prior to or during the study.
28. Close contact of anyone known to have COVID-19 infection within 30 days prior to vaccine administration.
29. Confirmed or suspected positive COVID-19 test results via diagnostic or antibody test.
30. Current treatment with investigational agents for prophylaxis of COVID-19.
31. Current use of any prescription or over-the-counter medications within 7 days prior to vaccination, unless approved by the investigator or necessary to manage a chronic condition.
32. Plans to travel outside the participating country from enrollment through 28 days after the second vaccination.
33. Healthcare worker at high risk of contracting SARS-CoV-2
34. Reside in a skilled nursing home, have a requirement for skilled nursing care, and/or non-ambulatory.
35. Medical or psychiatric condition including recent (with the past year) or active suicidal ideation/behavior or abnormality, self-reported or medically documented, that may increase the risk of study participation or make the participant inappropriate for the study based on the Investigator's judgement.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of 2-dose vaccination schedule of orally administered CoV2-OGEN1 by following local and systemic adverse events | Non serious AE are to assessed for 21-28 days after each study vaccination while serious AE are to be followed for atleast 6 months after completion of all study vaccinations
  Solicited local and systemic adverse events (may include Gi Disturbance)-Potential systemic events may include fever, fatigue, headache and chills following vaccination. Potential local events may include nausea, vomiting, diarrhea, and gastrointestinal discomfort following vaccination.

SECONDARY OUTCOMES:
To evaluate geometric mean fold rise (GMFR) | From baseline on day 43
  In mucosal IgA titer
To evaluate geometric mean fold rise (GMFR) | From baseline on day 43
  In serum IgG titer
To evaluate geometric mean fold rise (GMFR) | From baseline on day 43
  In serum IgA titer
To evaluate geometric mean titer (GMT) | On day 43
  Of mucosal antibody
To evaluate geometric mean titer (GMT) | On day 43
  Of serum antibody
To evaluate percentage of subjects | On day 43
  Seroconverted

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland Clinical Studies Ltd (NZCR OpCo Limited), Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No